CLINICAL TRIAL: NCT06146179
Title: Application Of Combined Anterior Suprascapular Nerve Block and Superficial Cervical Plexus Block In Reverse Shoulder Arthroplasty Surgery, A Case Series
Brief Title: Combined Anterior Suprascapular Nerve Block and Superficial Cervical Plexus Block In Shoulder Arthroplasty Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ebru Girgin Dinç, MD, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: 2023/0363
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Diaphragmatic Paralysis; Anterior Suprascapular Nerve Block; Superficial Cervical Plexus Block; Phrenic Nerve Paralysis
Keywords: diaphragmatic paralysis; anterior suprascapular nerve block; superficial cervical plexus block; reverse shoulder replacement; shoulder pain
MeSH Terms: conditions — Respiratory Paralysis; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Group 1: Combined Anterior Suprascapular Nerve Block and Superficial Cervical Plexus Block

SUMMARY:
The suprascapular nerve, originating from the C5 trunk, provides innervation to the acromioclavicular and glenohumeral joints. The supraclavicular nerve, a branch of the cervical plexus, contributes to the sensory innervation of the upper deltoid region. Cervical and brachial plexus blocks can cause diaphragm paralysis. This study examined the effects of low-volume combined anterior suprascapular nerve block and superficial cervical plexus block on pain and phrenic nerve in participants underwent reverse shoulder arthroplasty surgery.

DETAILED DESCRIPTION:
A retrospective analysis was performed on data obtained from eight participants who underwent reverse shoulder arthroplasty surgery. Anterior suprascapular nerve block and superficial cervical plexus block were applied to these participants. Anterior suprascapular nerve block was performed using 5 ml and superficial cervical plexus block was performed using 3 ml of %0,5 bupivacaine. Ultrasound was used to measure the diaphragm thickness at the end of inspiration and expiration, and to calculate the diaphragm thickness fraction. Postoperative pain management included patient-controlled analgesia with morphine, opioid consumption and VAS score recorded by pain observation forms.

Data will be collected by examining these pain observation forms and diaphragm thickness measurements.

ELIGIBILITY:
Inclusion Criteria:

* Population is defined by database within a given time frame
* Participants who underwent combined anterior suprascapular nerve block and superficial cervical plexus block in reverse shoulder arthroplasty surgery
* Participants aged 18-80
* ASA I-II-III

Exclusion Criteria:

* ASA score > III
* Pediatric individuals under 18 years of age
* Individuals who are pregnant
* Known diaphragmatic paralysis
* Had an allergy or toxicity to local anesthetic agents
* Have an opioid drug allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who underwent combined anterior suprascapular nerve block and superficial cervical plexus block in reverse shoulder arthroplasty surgery
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Change Ratio of Diaphragm Thickness Fraction | Postoperatively 30th. min.
  Postoperative Change Ratio of Diaphragm Thickness Fraction (%) at Postoperatively 30th. min.

SECONDARY OUTCOMES:
Pain Assessment with Visual Analogue Scale at postoperatively 30th. Min. | Postoperatively 30th. min
  Postoperative VAS score (Ranging from 0-10)
Pain Assessment with Visual Analogue Scale at postoperatively 4th. Hours. | Postoperatively 4th. hour
  Postoperative VAS score (Ranging from 0-10)
Pain Assessment with Visual Analogue Scale at postoperatively 6th. Hours. | Postoperatively 6th. hour
  Postoperative VAS score (Ranging from 0-10)
Pain Assessment with Visual Analogue Scale at postoperatively 12th. Hours. | Postoperatively 12th. hour
  Postoperative VAS score (Ranging from 0-10)
Pain Assessment with Visual Analogue Scale at postoperatively 24th. Hours. | Postoperatively 24th. hour
  Postoperative VAS score (Ranging from 0-10)
Opioid Consumption at postoperatively 30th. Min. | Postoperatively 30th. min.
  Postoperative Opioid Consumption with Morphine PCA (0.5 mg/cc, demand dose 2 cc, lock of time; 10 min. )
Opioid Consumption at postoperatively 4th. Hours. | Postoperatively 4th. hour
  Postoperative Opioid Consumption with Morphine PCA (0.5 mg/cc, demand dose 2 cc, lock of time; 10 min. )
Opioid Consumption at postoperatively 6th. Hours. | Postoperatively 6th. hour
  Postoperative Opioid Consumption with Morphine PCA (0.5 mg/cc, demand dose 2 cc, lock of time; 10 min. )
Opioid Consumption at postoperatively 12th. Hours. | Postoperatively 12th. hour
  Postoperative Opioid Consumption with Morphine PCA (0.5 mg/cc, demand dose 2 cc, lock of time; 10 min. )
Opioid Consumption at postoperatively 24th. Hours. | Postoperatively 24th. hour
  Postoperative Opioid Consumption with Morphine PCA (0.5 mg/cc, demand dose 2 cc, lock of time; 10 min. )

OTHER OUTCOMES:
Patient Satisfaction with 5 point Likert Patient Satisfaction scale at postoperatively 24th. Hours | Postoperatively 24th hour
  Postoperative 24th. hour 5 point Likert Patient Satisfaction scale (1-Very dissatisfied, 2 - Dissatisfied, 3 - Unsure, 4 - Satisfied, 5 - Very satisfied)
Postoperative Nausea and Vomiting | During Postoperatively 24 hour
  Postoperative Nausea and Vomiting Score ( PONV0: No Nausea, No vomiting; PONV1: Nausea present, No vomiting; PONV2: Nausea and vomiting present; PONV3: Vomiting>2 epizodes in 30th. min; PONV4:Vomiting>3 epizodes in 30th.min)

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Girgin Dinç, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No